## Statistical analysis plan Protocol 300A SITACLAMP

## Glucagon

- **1. Meal :**Comparison between the two groups are performed with parametric t-test for samples taken at -5, 15, 30, 45, 60, 90, 120 min
- 2. **Clamp.** Change in glucagon during the clamp, i.e., between min 150 and 210 are performed and comparison between the groups are performed with parametric t-test.

## Insulin, C-peptid, GIP and GLP-1

Comparison between the two groups are performed with parametric t-test for samples taken at -5, 15, 30, 45, 60, 90, 120, 150, 180, 210 and 240 min

## Epinephrine, norepinephrine, PP and cortisol

Change in epinephrine, norepinephrine, PP and cortisol during the clamp, i.e., between min 150 and 210 are performed and comparison between the groups are performed with parametric t-test.

Lund, December 12, 2015

Bo Ahrén, Pl